CLINICAL TRIAL: NCT03523533
Title: Peripherally Inserted Internal Jugular Catheters: an Observational Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator Decision & not a clinical trial.
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Tony Yen, Associate Professor, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-116
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Intravenous Drug Usage

STUDY DESIGN:
Intervention Model Description: This is an observational study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripherally-inserted internal jugular catheter (Experimental): All enrolled patients will receive a peripheral angiocatheter in the internal jugular vein, under dynamic ultrasound guidance.
  Interventions: Procedure: Angiocatheter

INTERVENTIONS:
Procedure: Angiocatheter — Placement of angiocatheter in internal jugular vein

SUMMARY:
This is an observational study intended to characterize the time-to-placement of peripherally-inserted internal jugular (PIJ) catheters in appropriate patients. As secondary outcomes and to ensure patient safety, the investigators will record and evaluate adverse outcomes, but the study is not powered to detect rare events.

DETAILED DESCRIPTION:
This is an observational study with one arm. All enrolled patients will receive a peripheral angiocatheter in the internal jugular vein. Approximately 60 subjects will be enrolled.

After recruitment and consent, an investigator will place the peripherally-inserted jugular (PIJ) catheters for this study, under ultrasound guidance. Clean technique similar to that used for traditional peripheral intravenous catheters will be used, including chlorhexidine skin preparation, caps, and sterile ultrasound gel with sterile occlusive dressing over the ultrasound transducer. For patients included in this study because of a clinically-determined need for a second IV line, the catheter will be placed after anesthesia induction. Patients included because of difficult IV access will have the PIJ catheter placed prior to induction.

The size of the angiocatheter will be left to the clinical discretion of the investigator, from among these choices: 18G x 2.5 inches, 16G x 2 inches, or 14G x 2 inches. All angiocatheters will be radiopaque in order to permit visualization in the event of any required imaging. Catheters will be placed with visualization under dynamic ultrasonography using a Sonosite S-Nerve ultrasound machine with 13-6 MHz 25 mm linear array. All catheters and ultrasound components are being used in accordance with their labeling.

The depth of catheter insertion into the internal jugular vein will be determined, and the catheter will be removed/replaced immediately if it is found to extend less than 1.0 cm into the vessel. If the catheter is removed or replaced, routine care will be followed: pressure will be held until bleeding subsides and the site dressed appropriately (e.g. gauze with tape or adhesive bandage). No more than three attempts will be made before abandoning the effort to place a PIJ catheter.

The PIJ catheter will be secured as per normal practice, with an adhesive IV securing device and an occlusive bandage placed over both the IV and its securing device.

The PIJ catheter will be used as usual during surgery. It will not be used for total parenteral nutrition or other continuous nutrient infusions.

In most cases, the PIJ catheter will be removed as usual before the patient is transferred to the floor, intensive care unit, or discharged home. In some cases, however, an appropriately authorized clinician may determine that the PIJ catheter should remain in place longer. If extended use of the PIJ catheter is indicated, it will be removed when it is either replaced as appropriate by another intravenous line or no longer needed.

Procedural data will be gathered on the day of surgery, and chart review will occur after surgery in order to capture any IV-related complications within the first week that were not immediately apparent.

ELIGIBILITY:
Inclusion Criteria: Adult elective-surgery patients at University of New Mexico Hospital main operating rooms, who do not require central venous catheters, and who either:

1. require a second intravenous access line (IV) as determined by the anesthesiologist, *or*
2. require a primary IV *and* are determined by the anesthesiologist to have difficult IV access, defined as two or more failed attempts at peripheral IV placement, in the absence of an indication for a central venous catheter.

Exclusion Criteria:

* Infection over the intended peripheral angiocatheter insertion site
* Cervical spine injury or instability
* Known abnormal neck anatomy
* Pregnancy
* Prisoners
* Clinical indication for central venous catheter
* Any pre-existing suspicion for bacteremia
* Adults unable to consent, as determined by ability to provide consent for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Yen, MD, Principal Investigator — University of New Mexico Health Sciences Center (HSC)
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peripherally-inserted Internal Jugular Catheter
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Peripherally-inserted Internal Jugular Catheter
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Catheter Placement Time
Description: Elapsed time from first contact of skin prep solution to completely secured/covered catheter
Time Frame: No more than 20 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Peripherally-inserted Internal Jugular Catheter
Number analyzed (Participants) | 5
minutes | 5.06 (0.78)

2. Secondary Outcome: Location of Insertion
Description: Choice of placement on patient's right or left side
Time Frame: No more than 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Peripherally-inserted Internal Jugular Catheter
Number analyzed (Participants) | 5
Participants
  Catheter placed on patient's right side | 5
  Catheter placed on patient's left side | 0

3. Secondary Outcome: Depth of Insertion
Description: Depth of catheter insertion in target blood vessel
Time Frame: No more than 20 minutes
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Peripherally-inserted Internal Jugular Catheter
Number analyzed (Participants) | 5
centimeters | 3.4 (1.2)

4. Secondary Outcome: Number of Attempts
Description: Count of attempts to successfully place catheter
Time Frame: No more than 20 minutes
Measure: Mean (Full Range); unit: Attempt
Arm/Group | Peripherally-inserted Internal Jugular Catheter
Number analyzed (Participants) | 5
Attempt | 1 [1 to 1]

5. Secondary Outcome: Number of Participants Experiencing Catheter-related Complications
Description: Count of subjects experiencing complications that are related to catheter placement
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Peripherally-inserted Internal Jugular Catheter
Number analyzed (Participants) | 5
Participants
  Patients experiencing carotid puncture | 0
  Patients experiencing pneumothorax | 0
  Patients experiencing thrombosis | 0
  Patients experiencing unexpectedly severe pain on placement | 0
  Patients experiencing hematoma | 0
  Patients experiencing injection-site infection | 0
  Patients experiencing none of these complications | 5

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | Peripherally-inserted Internal Jugular Catheter
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripherally-inserted Internal Jugular Catheter (N=5)
Loss of Catheter Patency (Product Issues) | 2 (2) — Loss of patency (open catheter allowing appropriate fluid flow)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03523533/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03523533/ICF_001.pdf